CLINICAL TRIAL: NCT05905926
Title: An Open-Label Long-Term Safety Study of Tenapanor for the Treatment of Irritable Bowel Syndrome With Constipation (IBS-C) in Pediatric Patients 6 to Less Than 18 Years Old
Brief Title: Safety Study of Tenapanor for the Treatment of Pediatric Patients (6 to Less Than 18 Years Old) With IBS-C
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TEN-01-306
Record Dates: First submitted 2023-03-07; First posted 2023-06-15 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome With Constipation (IBS-C)
MeSH Terms: interventions — tenapanor

STUDY DESIGN:
Intervention Model Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tenapanor (Experimental): Eligible patients from the parent study will continue tenapanor at the same dose assigned in the parent study which can be titrated to either 50 mg BID or 25 mg BID per Investigator guidance after a patient's first week on the assigned dose.
  Interventions: Drug: Tenapanor

INTERVENTIONS:
Drug: Tenapanor — Eligible patients from the parent study will continue tenapanor at the same dose assigned in the parent study. Doses can be titrated to either 50 mg BID or 25 mg BID
  Other Names: Ibsrela

SUMMARY:
Open-label long-term safety study of tenapanor in pediatric patients with IBS-C.

DETAILED DESCRIPTION:
Open-label long-term safety study of tenapanor in pediatric patients with IBS-C. Eligible patients who complete the parent study will have an option to enroll in this study.

Patients from the parent study will continue tenapanor at the same dose assigned in the parent study which can be titrated to either 50 mg BID or 25 mg BID per guidance in protocol after a patient's first week on the assigned dose. Patients will also return for study visits approximately every 6 weeks for safety assessments.

ELIGIBILITY:
Inclusion Criteria:

1. ≥6 and <18 years old at enrollment of either parent study
2. Patient completed the parent study immediately with adequate compliance with study procedures in the opinion of the Investigator
3. Females of child-bearing potential must have negative pregnancy test at the last visit of the parent study and confirm the use of appropriate contraception (including abstinence).
4. Subject is ambulatory
5. Written informed consent by parent/guardian/ Legally Authorized Representative (LAR) and a willingness of both subject and parent/guardian/LAR to participate in the study as it is described

Exclusion Criteria:

1. Patient discontinued prematurely from the parent study.
2. Any surgery on the stomach, small intestine or colon, excluding appendectomy or cholecystectomy
3. Pregnant or lactating women
4. If, in the opinion of the Investigator, patient is unable or unwilling to fulfill the requirements of the protocol

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Safety Measure Assessment (Adverse Event) | 40 weeks
  Incidence of AEs, SAEs and drug related adverse events
Safety Measure Assessment (ECG) | 40 weeks
  Descriptive summaries of ECG parameters (heart rate, PR-interval, QRS-duration, QT-interval, QTc-interval, and RR-interval)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Edelstein, PhD, Study Director — Ardelyx
Locations (22):
- United States (22):
  - G & L Research, LLC, Foley, Alabama
  - Advanced Research Center, Inc., Anaheim, California
  - Prohealth Research Center, Doral, Florida
  - I.H.S. Health, LLC, Kissimmee, Florida
  - Valencia Medical and Research Center, Miami, Florida
  - Florida Pharmaceutical Research and Associates, Inc., South Miami, Florida
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Mankato Clinic/ Javara Research Ltd, Mankato, Minnesota
  - Boys Town National Research Hospital, Boys Town, Nebraska
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Advantage Clinical Trials, The Bronx, New York
  - Atrium Health, Charlotte, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Prisma Health Children's Hospital, Greenville, South Carolina
  - Maspons Pediatric Gastro, El Paso, Texas
  - Texas Digestive Specialists, Harlingen, Texas
  - AIM Trials, LLC, Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Pioneer Research Solutions Inc, Sugar Land, Texas
  - Frontier Clinical Research, Kingwood, West Virginia